CLINICAL TRIAL: NCT05086172
Title: Ultrabrief Behavioral Activation for Reducing Alcohol Use
Acronym: UBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1369
Record Dates: First submitted 2021-09-24; First posted 2021-10-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Use Disorder, Mild; Alcohol Use Disorder, Moderate
MeSH Terms: conditions — Alcoholism; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This is an early pilot study that will compare an interventional assignment group to an "assessment only" control. The focus is on feasibility and acceptance of such a short intervention. The intervention is an ultrabrief, single-session (90 minute) administration of UBA, a psychotherapy intervention derived from the evidence-based LETS ACT Behavioral Activation treatment for substance use disorder. However, the investigators will also measure the difference of change in alcohol use behavior between groups as an additional outcome to gain an initial understanding of the magnitude of the effect for the design of future controlled studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UBA Arm (Experimental): All subjects in this arm will receive ultrabrief behavioral activation therapy via a single, 90-minute session.
  Interventions: Behavioral: Ultrabrief Behavioral Activation
- Control Arm (No Intervention): All subjects in this arm will complete all study assessment instruments collected in the interventional arm but will not receive an intervention.

INTERVENTIONS:
Behavioral: Ultrabrief Behavioral Activation — The ultrabrief behavior activation (UBA) intervention is a condensed version of the LETS ACT intervention. The main treatment elements include: (1) explanation of treatment rationale to facilitate behavior change via increased engagement in values-related activities, (2) identification of participant-specific values via detailed assessment of life areas, values and activities, (3) values-based activity planning and scheduling, and (4) post-treatment planning. The overall goal of behavioral activation (BA) is to shift from values-incongruent behavior (including alcohol use) to behaviors that provide positive reinforcement and environmental reward with the overall goal of increasing the number of engaged-in, value-based activities. This intervention will take 90 minutes.
  Other Names: UBA
  Arms: UBA Arm

SUMMARY:
This is a pilot study to assess feasibility, acceptability, and preliminary efficacy of a single-session ("ultrabrief") psychological intervention to reduce alcohol use in participants with mild to moderate alcohol use disorder (AUD). The intervention is a condensed form of the Life Enhancement Treatment for Substance Use (LETS ACT), behavioral activation (BA) for co-morbid depression and substance use. The investigators hypothesize that UBA is feasible and acceptable. The investigators hypothesize that UBA will reduce overall total alcohol consumption as determined by self-report measures capturing drinking behavior for the 3 months prior to treatment versus the 3 months after treatment when compared to an "assessment only" condition.

DETAILED DESCRIPTION:
This is a pilot study to investigate feasibility, acceptability, and preliminary efficacy of an ultrabrief behavioral activation (UBA) intervention for people with a mild to moderate alcohol use disorder. UBA is a psychotherapy intervention derived from the evidence-based LETS ACT BA treatment for substance use disorder. All clinical interviews and the UBA intervention itself will be audio recorded for the purposes of training and to determine reliability and adherence to diagnostic and treatment protocols. No biological samples or signals are collected in this study. The study comprises a phone screening for eligibility, three in-person study visits (initial baseline assessment (BL), UBA intervention session, and 2-week post-treatment assessment) and two follow up phone call assessments (1 month and 3 months after treatment completion). There will be an "assessment only" study arm that will act as a control group which mirrors all aspects of the intervention arm except the "assessment only" arm will receive no intervention. The ultrabrief behavior activation (UBA) intervention is a condensed version of the LETS ACT intervention. The main treatment elements include: (1) explanation of treatment rationale to facilitate behavior change via increased engagement in values-related activities, (2) identification of participant-specific values via detailed assessment of life areas, values and activities, (3) values-based activity planning and scheduling, and (4) post-treatment planning. The overall goal of BA is to shift from values-incongruent behavior (including alcohol use) to behaviors that provide positive reinforcement and environmental reward with the overall goal of increasing the number of engaged-in, value-based activities. This intervention will take 90 minutes. Following intervention completion, therapists will complete a therapist questionnaire and participants will schedule follow-up assessments to occur 2-weeks, 1-month, and 3-months post-treatment. There will be three follow-up contacts with study participants, one in-person visit occurring 2 weeks after the UBA intervention and two phone-based assessments occurring 1 and 3 months following treatment respectively. Follow-up 1 focuses on the treatment experience whereas Follow-up 2 and 3 focus on change in alcohol use and related behaviors and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild or moderate alcohol use disorder based on Diagnostic and Statistical Manual-V (DSM-5) criteria
* Age: 18 years or older

Exclusion Criteria:

* Psychotic disorder as determined by the Mini-International Neuropsychiatric Interview (MINI)
* Current suicidality as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Diagnosis of severe alcohol or substance use disorder (AUD;SUD) based on MINI
* Receiving concurrent psychotherapy for a mental health-related condition
* Concurrent use of FDA approved medications for the treatment of a substance us disorder
* Change in psychiatric medication in the last four weeks
* The inability to give informed, voluntary, written consent to participate
* Inability to communicate effectively in English as determined by interaction with study personnel
* Anything else that in the assessment of the investigational team is not conducive to successful completion of study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Feasibility via average rate of enrollment of eligible participants | Through completion of the study, an average of 1 year
  The investigators will compute the average rate of enrollment of eligible participants when 20 participants have concluded study participation to determine the feasibility of such interventions.
Feasibility via computed fraction of participants who have completed all assessment in this study | Baseline up to 3-months Post treatment (Follow up 3)
  The investigators will compute the fraction of participants who have completed all assessments in this study (baseline, 2-weeks post treatment, 1-month post treatment-3-months post treatment)
Acceptability via summary scores and statistics of study-designed treatment engagement and acceptability assessment instruments | 2 weeks Post Treatment (2 week follow-up)
  Acceptability will be characterized by computing summary scores and their corresponding statistics from the Treatment Engagement and Acceptability Assessment (TEA) designed for this study. Scores on the TEA range from a minimum score of 20 to a maximum score of 100, with higher scores indicating greater treatment engagement and acceptability.

SECONDARY OUTCOMES:
Change in alcohol consumption via average amount of alcohol consumed per drinking day | 3 months prior to Baseline up to 3-months post treatment
  The investigators will compute the change in total alcohol consumption from the three months prior to Baseline up to 3 months post treatment based on the average amount of alcohol consumed per drinking day in the 3 months prior to baseline compared to the average amount of alcohol consumed per drinking day reported in the 3 months post treatment as recorded on the time-line followback (TLFB) in both study arms and assess a pre-treatment, post-treatment difference between groups.
Change in alcohol consumption via number of drinking days | 3 months prior to Baseline up to 3-months post treatment
  The investigators will compute the change in total alcohol consumption from the three months prior to Baseline up to 3 months post treatment based on the number of reported drinking days in the 3 months prior to baseline compared to the number of drinking days reported in the 3 months post treatment as recorded on the time-line followback (TLFB) in both study arms and assess a pre-treatment, post-treatment difference between groups.
Feasibility via computed fraction of participants that successfully completed at least 1 of each activity independently as per record in treatment booklet | 2 weeks Post treatment
  The investigators will compute the fraction of participants who filled in the treatment booklets in a way that the participants completed at least one of each activity independently at-home (i.e., at least 1 activity and value for at least 3 life areas AND at least 2 alternative activities to alcohol AND at least 1 activity daily for 14 days). This measures feasibility of participants performing work that would be done in-session in longer interventions at home on their own for UBA.
Feasibility via the therapist questionnaire (TQ) developed by the investigators for this study | Immediately following Treatment Session
  The investigators will assemble formal feedback from the form for the therapist to fill out (TQ); 3 sub-scores for material covered, acceptance by participant, and participant engagement. The Material Covered subscale ranges from a minimum score of 0 to a maximum score of 10, with higher scores indicating less thorough material coverage. The Acceptance sub-scale ranges from a minimum score of 4 to a maximum score of 20, with higher scores indicating higher levels of acceptance. The Participant Engagement sub-scale ranges from a minimum score of 5 to a maximum score of 25, with higher scores indicating higher levels of participant engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Daughters, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after de-identification.
Time Frame: Immediately following publication without expiry.
Access Criteria: Researchers requesting the use of the provided de-identified data should direct inquiries to Stacey Daughters (daughter@unc.edu) and should have received approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.

REFERENCES:
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Babor TF, Del Boca F, Bray JW. Screening, Brief Intervention and Referral to Treatment: implications of SAMHSA's SBIRT initiative for substance abuse policy and practice. Addiction. 2017 Feb;112 Suppl 2:110-117. doi: 10.1111/add.13675. PMID 28074569
- [Background] Miller WR, Wilbourne PL. Mesa Grande: a methodological analysis of clinical trials of treatments for alcohol use disorders. Addiction. 2002 Mar;97(3):265-77. doi: 10.1046/j.1360-0443.2002.00019.x. PMID 11964100
- [Background] Gawrysiak, M., C. Nicholas, and D.R. Hopko, Behavioral activation for moderately depressed university students: Randomized controlled trial. Journal of Counseling Psychology, 2009. 56(3): p. 468-475.
- [Background] Parra, P.A.R., J.I. Uribe, and J.M. Bianchi, Effectiveness of a Single Session Protocol of Behavioral Activation in College Students with Depressive Symptomatology. International journal of psychology and psychological therapy, 2019. 19(1): p. 5-14
- [Background] Daughters SB, Magidson JF, Anand D, Seitz-Brown CJ, Chen Y, Baker S. The effect of a behavioral activation treatment for substance use on post-treatment abstinence: a randomized controlled trial. Addiction. 2018 Mar;113(3):535-544. doi: 10.1111/add.14049. Epub 2017 Nov 19. PMID 28963853
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Blanchard KA, Morgenstern J, Morgan TJ, Lobouvie EW, Bux DA. Assessing consequences of substance use: psychometric properties of the inventory of drug use consequences. Psychol Addict Behav. 2003 Dec;17(4):328-31. doi: 10.1037/0893-164X.17.4.328. PMID 14640829
- [Background] Carver, C. S., & White, T. L. (1994). Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS scales. Journal of Personality and Social Psychology, 67, 319-333
- [Background] Carvalho JP, Gawrysiak MJ, Hellmuth JC, McNulty JK, Magidson JF, Lejuez CW, Hopko DR. The reward probability index: design and validation of a scale measuring access to environmental reward. Behav Ther. 2011 Jun;42(2):249-62. doi: 10.1016/j.beth.2010.05.004. Epub 2011 Jan 18. PMID 21496510
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] First, M. B., Gibbon, M., Spitzer, R. L., Williams, J. B. W., & Benjamin, L. S. (1997). Structured Clinical Interview for DSM-IV Axis II personality disorders (SCID-II). Washington, DC: American Psychiatric Press.
- [Background] Hatcher, R. L., & Gillaspy, J. A. (2006). Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy Research, 16(1), 12-25. https://doi.org/10.1080/10503300500352500
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Jastak, S., & Wilkinson Gary, W. (1984). The Wide Range Achievement Test-revised, WRAT-R. Jastak Associates.
- [Background] Kanter, J. W., Mulick, P. S., Busch, A. M., Berlin, K. S., & Martell, C. R. (2007). The Behavioral Activation for Depression Scale (BADS): Psychometric properties and factor structure. Journal of Psychopathology and Behavioral Assessment, 29(3), 191-202. https://doi.org/10.1007/s10862-006-9038-5
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] McNeely J, Wu LT, Subramaniam G, Sharma G, Cathers LA, Svikis D, Sleiter L, Russell L, Nordeck C, Sharma A, O'Grady KE, Bouk LB, Cushing C, King J, Wahle A, Schwartz RP. Performance of the Tobacco, Alcohol, Prescription Medication, and Other Substance Use (TAPS) Tool for Substance Use Screening in Primary Care Patients. Ann Intern Med. 2016 Nov 15;165(10):690-699. doi: 10.7326/M16-0317. Epub 2016 Sep 6. PMID 27595276
- [Background] Miller, W. R., & Tonigan, J. S. (1996). Assessing drinkers' motivation for change: The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). Psychology of Addictive Behaviors, 10(2), 81-89. https://doi.org/10.1037/0893-164X.10.2.81
- [Background] Posner, K., Brent, D., Lucas, C., Gould, M., Stanley, B., Brown, G., ... & Mann, J. (2008). Columbia-suicide severity rating scale (C-SSRS). New York, NY: Columbia University Medical Center, 10.
- [Background] Sheehan, D. V., Lecrubier, Y., Janavs, J., Baker, N., Harnett Sheehan, K., Knapp, E., ... & Lepine, J. P. (2016). Mini International Neuropsychiatric Interview English version 7.0. 2 for DSM-5. University of South Florida College of Medicine.
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Sobell LC, Maisto SA, Sobell MB, Cooper AM. Reliability of alcohol abusers' self-reports of drinking behavior. Behav Res Ther. 1979;17(2):157-60. doi: 10.1016/0005-7967(79)90025-1. No abstract available. PMID 426744
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404
- [Background] Wilson, K. G., Sandoz, E. K., Kitchens, J., & Roberts, M. (2010). The Valued Living Questionnaire: Defining and measuring valued action within a behavioral framework. The Psychological Record, 60(2), 249-272.
- See also: Co-Investigator's Lab Website — http://www.frohlichlab.org/
- See also: Study Research for Me with study information and links for interested individuals — http://STUDIES.UNC.EDU/21-1369